CLINICAL TRIAL: NCT02034409
Title: A Pilot Trial to Assess Low-Intensity Ultrasound in Osteoarthritis
Acronym: PLUS+OA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-006-13S; CXI01CX000954-01A1 (Other: eRA project Reference)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Degenerative
Keywords: Knee Osteoarthritis; Pulsed Low Intensity Ultrasound
MeSH Terms: conditions — Joint Diseases; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants in this double-blind, randomized, sham-controlled trial will be randomly assigned to receive either sham or PLIUS device for 48 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham (Sham Comparator): Treatment to index knee with sham device for 48 weeks
  Interventions: Device: Sham Comparator
- PLIUS (Experimental): Treatment to index knee with PLIUS device for 48 weeks
  Interventions: Device: Pulsed Low Intensity Ultrasound

INTERVENTIONS:
Device: Pulsed Low Intensity Ultrasound — 20 minutes daily for 48 weeks
  Arms: PLIUS
Device: Sham Comparator — 20 minutes daily for 48 weeks
  Arms: Sham

SUMMARY:
The purpose of this exploratory trial is to investigate whether PLIUS is potentially effective as a disease and symptom modifying intervention in patients with early knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA), the most common form of arthritis, is a prevalent and debilitating disease without therapies that alter disease progress and is currently managed with symptom-modifying therapies that are only modestly effective. In spite of substantial progress in understanding the pathogenesis of OA, no effective disease modifying interventions have been established. Degenerative joint cartilage is a central feature of OA, yet joint cartilage has a limited capacity for repair. Results from animal research demonstrate that pulsed low intensity ultrasound (PLIUS) mechanically stimulates, and may promote, cartilage repair. This exploratory trial will investigate whether PLIUS is potentially effective as a disease and symptom modifying intervention in patients with early knee OA.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older, and a US Military Veteran
* Clinical symptoms of osteoarthritis for at least 6 months
* Pain in the index knee on motion or weight bearing for the majority of days during the month before screening
* Clinical diagnosis of primary osteoarthritis of the knee based on clinical and radiographic criteria
* American Rheumatism Association Functional Class I, II, or III
* Females of childbearing potential must be willing to use a reliable form of medically acceptable contraception

Exclusion Criteria:

* Concurrent medical/arthritis condition(s), or any other illness per the opinion of the investigator, that could interfere with the evaluation of pain or efficacy
* Spine or hip pain of significant magnitude
* History of significant ligament or meniscal injury of the index joint requiring surgical repair
* Arthroscopy of the index knee within 6 months of study entry
* Unable to undergo MRI of the knee
* Pregnancy or lactation
* Corticosteroid treatment within 1 to 3 months prior to study entry
* Intra-articular injection of hyaluronic acid or congeners to the index knee within 6 months of study entry
* Use of excluded therapy(ies) prior to study entry
* Use of disease modifying anti-rheumatic medications and chronic tetracycline or its derivatives
* Exposure to glucosamine, chondroitin sulfate, or any other investigational treatment, within 1 month of study entry
* Use of any medical therapy, complementary or alternative regimens for the treatment of osteoarthritis within 7 days prior to study entry
* Initiation of physical therapy or muscle conditioning program to the lower extremities within 2 months within 2 months prior to study entry
* Unlikely to comply with study requirements

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Clegg, MD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (3):
- United States (3):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sawitzke AD, Jackson CG, Carlson K, Bizien MD, Leiner M, Reda DJ, Sindowski T, Hanrahan C, Spencer RG, Kwoh CK, Lee SJ, Hose K, Robin L, Cain DW, Taylor MD, Bangerter N, Finco M, Clegg DO. Effect of Pulsed Low-Intensity Ultrasonography on Symptom Relief and Tibiofemoral Articular Cartilage Thickness Among Veterans Affairs Enrollees With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e220632. doi: 10.1001/jamanetworkopen.2022.0632. PMID 35258579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 2 medical centers between May 2015 and January 2019. The first participant was enrolled May 2017 and the last participant was enrolled in January 2019.
Pre-assignment Details: 140 participants began, and 136 completed, the 4-Week Sham Run-in Period. 4 of the 140 Sham Run-in participants were withdrawn due to being less than 80% treatment compliance.
Groups:
- Sham: Treatment to index knee with sham device for 48 weeks
  ShamComparator: 20 minutes daily for 48 weeks
- PLIUS (Pulsed Low Intensity UltraSound): Treatment to index knee with PLIUS device for 48 weeks
  PLIUS device: 20 minutes daily for 48 weeks
Period: Sham Run-in Period
Arm/Group | Sham | PLIUS (Pulsed Low Intensity UltraSound)
Started | 140 | 0 (Number started is zero because there is no PLIUS arm in Sham Run-in Period)
Completed | 136 | 0 (Number started is zero because there is no PLIUS arm in Sham Run-in Period)
Not Completed | 4 | 0
Not completed — Participants withdrawn per protocol because less than 80% treatment compliance | 4 | 0
Period: Sham-Controlled Treatment Period
Arm/Group | Sham | PLIUS (Pulsed Low Intensity UltraSound)
Started | 67 (Number started in Sham Arm of Sham-Controlled Treatment Period Milestone not equal to Sham Run-in Period Milestone because participants in this Milestone are randomly assigned to either Sham or PLIUS treatment arm.) | 69 (Number started in PLIUS Arm of Sham-Controlled Treatment Period Milestone not equal to Sham Run-in Period Milestone because participants in this Milestone are randomly assigned to either Sham or PLIUS treatment arm.)
Completed | 55 | 54
Not Completed | 12 | 15
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Physician Decision | 1 | 3
Not completed — misrandomized | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | PLIUS | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.9) | 62.9 (10.5) | 63.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 58 | 61 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 23
  Not Hispanic or Latino | 55 | 54 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 52 | 48 | 100
  More than one race | 3 | 9 | 12
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 67 | 132
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index Population: Needed data for baseline measure only available for 130 participants
  kg/m^2
    number analyzed (Participants) | 64 | 66 | 130
    (all) | 31.6 (5.5) | 31.8 (5.4) | 31.7 (5.5)
Years with Osteoarthritis [Mean (Standard Deviation); unit: years] — Participant reported duration of osteoarthritis
  years | 11.7 (11.2) | 15.0 (13.2) | 13.4 (12.3)
ARA Functional Class [Count of Participants; unit: Participants] — American Rheumatism Association (ARA) Functional Class categorize global functional capacity and is assessed by a qualified health professional. A higher class indicates a worsening of functional capacity.
  Class I - Completely able to perform usual activities of daily living. Class II - Able to perform usual self-care and vocational activities but limited in avocational activities.
  Class III - Able to perform usual self-care activities but limited in vocational and avocational activities.
  Class IV - Limited in ability to perform usual self-care, vocational, and avocational activities.
  Participants
    Class I | 0 | 2 | 2
    Class II | 48 | 52 | 100
    Class III | 17 | 13 | 30
    Class IV | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Measure: a) Symptom Reduction: OMERACT-OARSI Treatment Responsiveness
Description: Outcome Measures in Rheumatology Clinical Trials- Osteoarthritis Research Society International (OMERACT-OARSI) Response incorporates changes in pain and global assessment to define response in OA clinical trials. A response is classified as: 1) An improvement in either pain or function of at least 50 percent accompanied by an absolute decrease of at least 20 mm on the visual-analogue scale for pain or function, OR 2) The occurrence of at least two of the following: a) a decrease in pain of at least 20 percent accompanied by a decrease of at least 10 mm on the visual-analogue scale; b) an improvement in function of at least 20 percent and a decrease of at least 10 mm on the visual-analogue scale; c) an increase in the patient's global assessment score by at least 20 percent accompanied by a decrease of at least 10 mm on the visual-analogue scale
Time Frame: 48 weeks
Population: Participants with baseline and 48 week values.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 55 | 54
Participants
  OMERACT-OARSI responders | 37 | 38
  OMERACT-OARSI non-responders | 18 | 16
Statistical Analysis 1: Comparison: Sham vs PLIUS; Sample size has been calculated with ranking and selection methodology, a procedure used for Phase II trials. The purpose of the procedure as applied to this study is to identify whether PLIUS has a high probability of being more effective than sham. This is accomplished by obtaining sample estimates of the outcome for the PLIUS and sham groups and determining whether the PLIUS group outcome is better by the pre-specified margin of difference; Test type: Non-Inferiority — For the 48-week OMERACT-OARSI response the minimally clinically significant difference is an absolute rate difference of 10% between sham and PLIUS groups. With a total sample size of 144 the probability of correctly selecting the group with the greatest OORR is at least 0.885 assuming (δ=10%) that the sham group is drawn from a population with a 50% response rate and the PLIUS group is drawn from a population with response rate of at least 60% or at most 40%; Since the ranking and selection procedures are fundamentally different from traditional hypothesis testing, concepts of statistical significance and power have no direct analogue

2. Primary Outcome: Co-Primary Measure: b) Disease Modification as Measured by Change From Baseline in Cartilage Thickness of the Central Medial Femoral Condyle Disease
Description: The study has been designed to determine if PLIUS potentially diminishes articular cartilage thinning by measuring cartilage thickness in the tibial femoral joint. The measure selected to best evaluate this is cartilage thickness of the central medial femoral condyle because studies of the OAI (Osteoarthritis Initiative) data have shown this region to be among those most sensitive to change and, due to the anatomical positioning of the device, the most likely to be affected by treatment.
Time Frame: Baseline, 48 weeks
Population: Participants with baseline and 48 week value
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 50 | 48
μm | -42.2 (297.0) | -73.8 (168.1)
Statistical Analysis 1: Comparison: Sham vs PLIUS; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — For the 48-week cartilage change outcome measure the minimally clinically significant difference is 33 μm. With a difference of 33 μm, σ=152 μm standard deviation, k=2 groups, and P=0.90 probability to obtain τ=1.8124, which we use to estimate the per-group sample size: n=σ2(τ/δ*)2=72 or a total of 144; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in WOMAC Stiffness Subscale Score
Description: The WOMAC® Index questionnaire is a tri-dimensional, disease-specific, self-administered, health status measure. It probes clinically important, patient-relevant symptoms in the areas of pain, stiffness and physical function in patients with osteoarthritis of the hip and/or knee. The WOMAC has been linguistically validated and is a reliable and responsive measure of outcome, and has been used in diverse clinical and interventional environments. Range is from 0 - 200. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Change from Baseline to week 24 | -33.6 [-47.6 to -19.7] | -27.7 [-40.2 to -15.1]
  Change from Baseline to week 48 | -49.8 [-64.6 to -35.1] | -37.1 [-51.6 to -22.6]

4. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Score
Description: The WOMAC® Index questionnaire [33] is a tri-dimensional, disease-specific, self-administered, health status measure. It probes clinically important, patient-relevant symptoms in the areas of pain, stiffness and physical function in patients with osteoarthritis of the hip and/or knee. The WOMAC has been linguistically validated and is a reliable and responsive measure of outcome, and has been used in diverse clinical and interventional environments. WOMAC pain scores from 0-500 mm. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale mm
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale mm
  Change from Baseline to week 24 | -84.2 [-109.4 to -58.9] | -91.4 [-111.1 to -71.7]
  Change from Baseline to week 48 | -117.1 [-146.2 to -87.9] | -93.4 [-124.4 to -62.3]

5. Secondary Outcome: Change From Baseline in WOMAC Functional Limits Subscale Score
Description: The WOMAC® Index questionnaire [33] is a tri-dimensional, disease-specific, self-administered, health status measure. It probes clinically important, patient-relevant symptoms in the areas of pain, stiffness and physical function in patients with osteoarthritis of the hip and/or knee. The WOMAC has been linguistically validated and is a reliable and responsive measure of outcome, and has been used in diverse clinical and interventional environments. Range is from 0 - 1700. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Change from Baseline to week 24 | -285.2 [-377.1 to -193.2] | -241.1 [-316.9 to -165.4]
  Change from Baseline to week 48 | -407.3 [-510.8 to -303.7] | -283.1 [-399.7 to -166.5]

6. Secondary Outcome: Change From Baseline in Total WOMAC Score
Description: The WOMAC® Index questionnaire is a tri-dimensional, disease-specific, self-administered, health status measure. It probes clinically important, patient-relevant symptoms in the areas of pain, stiffness and physical function in patients with osteoarthritis of the hip and/or knee. The WOMAC has been linguistically validated and is a reliable and responsive measure of outcome, and has been used in diverse clinical and interventional environments. Range is from 0 - 2400. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Change from Baseline to week 24 | -403.0 [-527.3 to -278.6] | -360.2 [-460.8 to -259.5]
  Change from Baseline to week 48 | -574.1 [-713.8 to -434.4] | -413.6 [-571.4 to -255.7]

7. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Status
Description: A patient global assessment of disease status on a Visual Analog Scale (VAS) will be measured at each clinic visit. Patients will be asked to quantify their disease status on a 100 mm VAS as follows: "Considering all the ways your arthritis of the knee affects you, mark 'X' on the scale for how well you are doing." The scale shows the left hand marker "Very Well", and the right hand marker "Very Poor." Range 0 to 100 mm. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Change from Baseline to Week 24 | -16.6 [-23.3 to -9.9] | -15.0 [-21.4 to -8.7]
  Change from Baseline to Week 48 | -23.7 [-30.8 to -16.5] | -17.6 [-26.3 to -9.0]

8. Secondary Outcome: Change From Baseline in Investigator Global Assessment of Disease Status
Description: An investigator global assessment of disease status on a 100 mm VAS was measured at each clinic visit as follows: "Make a global assessment of the patient's disease status, with regard to the index knee, by marking an 'X' on the scale below.", with left hand marker "Very Well" and right hand marker "Very Poor." Range 0 to 100 mm. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Change from Baseline to Week 24 | -18.4 [-25.0 to -11.9] | -15.8 [-22.5 to -9.0]
  Change from Baseline to Week 48 | -28.6 [-36.6 to -20.6] | -18.9 [-27.9 to -9.9]

9. Secondary Outcome: Change From Baseline in Intermittent and Constant Osteoarthritis Pain (ICOAP) Constant Pain Subscale
Description: This 11-item tool is designed to assess pain in individuals with knee osteoarthritis taking into account both constant and intermittent pain experiences. This tool is designed to be interviewer-administered. Study participants are asked to respond to the questionnaire items based on index knee in the past week (i.e., past 7-day period). Study participants responded to all questions for the same joint. This tool is intended to be responsive to change in OA pain over time or with treatment. Range 0 to 100 mm. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent To Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Change from Baseline to Week 24 | -14.6 [-20.1 to 9.1] | -12.4 [-18.0 to -6.8]
  Change from Baseline to Week 48 | -18.4 [-24.0 to -12.8] | -13.7 [-20.7 to -6.7]

10. Secondary Outcome: Change From Baseline in Intermittent and Constant Osteoarthritis Pain (ICOAP) Intermittent Pain Subscale
Description: This 11-item tool is designed to assess pain in individuals with knee osteoarthritis taking into account both constant and intermittent pain experiences. This tool is designed to be interviewer-administered and takes less than 10 minutes to complete. Study participants will be asked to respond to the questionnaire items based on index knee in the past week (i.e., past 7-day period). Study participants will respond to all questions for the same joint. This tool is intended to be responsive to change in OA pain over time or with treatment. Range 0 to 100 mm. The higher the score, the worse the symptoms.
Time Frame: Baseline, week 24, week 48
Population: Intent To Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Baseline to Week 24 | -17.7 [-23.2 to -12.3] | -13.4 [-18.2 to -8.5]
  Baseline to Week 48 | -20.2 [-26.8 to -13.6] | -15.0 [-21.5 to -8.5]

11. Secondary Outcome: Change From Baseline in Intermittent and Constant Osteoarthritis Pain (ICOAP) Total Pain Score
Description: as for outcome 10
Time Frame: Baseline, week 24, week 48
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Visual Analog Scale (mm)
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
Visual Analog Scale (mm)
  Change from Baseline to Week 24 | -16.3 [-21.3 to -11.3] | -12.9 [-17.9 to -8.0]
  Change from Baseline to Week 48 | -19.4 [-25.2 to 13.6] | -14.4 [-20.8 to -7.9]

12. Secondary Outcome: Number of Participants Discontinuing the Study Device Due to an Adverse Device Event
Description: Difference between study groups in number of participants who discontinued usage of the study device due to adverse device events at 4, 8, 12, 24, 36, and 48-week visits.
Time Frame: Baseline, 4, 8, 12, 24, 36, and 48-week visits
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | Sham | PLIUS
Number analyzed (Participants) | 65 | 67
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 48 weeks.
Arm/Group | Sham | PLIUS
All-Cause Mortality (participants affected / at risk) | 1/65 | 0/67
Serious Adverse Events (participants affected / at risk) | 13/65 | 19/67
Other Adverse Events (participants affected / at risk) | 0/65 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=65) | PLIUS (N=67)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angina, Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block, complete (Cardiac disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Dural arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lipoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Prostatectomy (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Infections and infestations) | 0 (0) | 1 (1)
Shoulder arthroplasty (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal laminectomy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02034409/Prot_SAP_000.pdf